CLINICAL TRIAL: NCT02178280
Title: Phase 1 Study of Liver Transplantation Combined With Neoadjuvant Radiochemotherapy for Unresectable Hilar Cholangiocarcinoma
Brief Title: Safety Study of Liver Transplantation for Hilar Cholangiocarcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Ding Yitao, Nanjing DrumTower Hospital, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20140615
Record Dates: First submitted 2014-06-14; First posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Hilar Cholangiocarcinoma
MeSH Terms: conditions — Klatskin Tumor | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- unresectable hilar cholangiocarcinoma (No Intervention): control group
- liver transplantation (Experimental): liver transplantation combined with neoadjuvant radiochemotherapy
  Interventions: Other: liver transplantation combined with neoadjuvant therapy

INTERVENTIONS:
Other: liver transplantation combined with neoadjuvant therapy — liver transplantation combined with neoadjuvant radiochemotherapy
  Arms: liver transplantation

SUMMARY:
Hilar cholangiocarcinoma is a highly malignant tumor. Surgical resection or simple liver transplantation leads to poor prognosis accompanied by high recurrence rate and low survival rate. The newly proposed neoadjuvant therapy with liver transplantation strategy shows promising clinical application, which once reported 5-year survival rate 82%. However, transplantation centers conducting this kind of research are limited due to its complexity and long-term. The investigators would like to conduct a clinical trial for only unresectable hilar cholangiocarcinoma patients who should take neoadjuvant brachytherapy and chemoradiotherapy followed by orthotopic liver transplantation.

DETAILED DESCRIPTION:
The enrolled patients should be prescribed with several examinations when admitted to hospital consisting of CT, MRI, MRCP, ECT, PET/CT and other laboratory tests. All preoperative examinations must indicate that enrolled individuals should be diagnosed as unresectable hilar cholangiocarcinoma. In addition, repetitive ERCP manipulations are needed in order to obtain positive results by brush cytology. Of course, all enrolled patients should be adherent to the fundamental principles of liver transplantation.

We employed I-125 radioactive plastic stents (patent No: ZL 201610116321.3) to conduct brachytherapy. Each stent composed of a drainage tube with a stab at both ends that had a stabilizing effect. Two opposite channels were made in the wall of stents paralleling the drainage lumen, with irradiation window in the lateral wall of the channel. The diameter of the channel is a bit smaller than that of the radioactive seeds, so as is the length and width of irradiation windows. The stents are so designed to immobilize seeds and radiate properly. The radioactive I-125 seeds were 4.5 mm long and 0.8 mm thick, and their half-life was 60.1 days. The nasobiliary radiography was performed to determine the length of involvement of bile duct.Corresponding radioactive seeds are then put in appropriate location with biliary stents by ERCP procedure.

About a month later, external beam radiotherapy was administrated to a target dose of 30Gy in 30 fractions, 1.5Gy twice per day. Concomitantly, Intravenous capecitabine was given at 1.0g bid for two weeks, which is repeated after 14 days until transplantation.

Immunosuppressive therapy was provided with tacrolimus, mycophenolate and corticosteroids. Corticosteroids were withdrawn a week later. Chemotherapy was continued 1 month after OLT with expected 3 courses.

ELIGIBILITY:
Inclusion Criteria:

unresectable hilar cholangiocarcinoma tumor diameter less than 3 cm adherence to liver transplantation requirements

Exclusion Criteria:

intrahepatic cholangiocarcinoma uncontrolled infection intrahepatic or extrahepatic metastasis distant lymph node metastasis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
survival rate | 1-yr survival rate
survival rate | 3-yr survival rate
survival rate | 5-yr survival rate
tumor-free survival rate | 1-yr tumor-free survival rate
tumor-free survival rate | 3-yr tumor-free survival rate
tumor-free survival rate | 5-yr tumor-free survival rate

SECONDARY OUTCOMES:
acute rejection rate | usually within 2 months after liver transplantation
chronic rejection rate | usually 2 months upon liver transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Yitao Ding, Study Chair — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Hepatobiliary department, Nanjing DrumTower Hospital, Nanjing, Jiangsu, China